CLINICAL TRIAL: NCT00943007
Title: Randomized Assessment of Conventional Neuronavigation Versus Intraoperative MRI for the Neurosurgical Treatment of Glioblastomas
Brief Title: Comparison of Standard Neuronavigation With Intraoperative Magnetic Resonance Imaging (MRI) for the Neurosurgical Treatment of Malignant Brain Tumors
Acronym: RACING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MEC 08-2-055
Record Dates: First submitted 2009-07-20; First posted 2009-07-21 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional Neuronavigation (Active Comparator): Standard form of neuronavigation: based on preoperative MRI without intraoperative correction for brain shift
  Interventions: Device: Stealth Station
- Intraoperative MRI (Experimental): Standard neuronavigation plus intraoperative MRI to correct for brain shift
  Interventions: Device: PoleStar N20

INTERVENTIONS:
Device: Stealth Station — Neuronavigation based on preoperative MRI
  Other Names: cNN
  Arms: Conventional Neuronavigation
Device: PoleStar N20 — Intraoperative MRI guided surgery
  Other Names: iMRI
  Arms: Intraoperative MRI

SUMMARY:
The treatment of a specific subtype of highly malignant brain tumor (called "glioblastoma" or "glioblastoma multiforme") consists of neurosurgical resection, followed by radiotherapy and mostly chemotherapy as well. Increased extent of tumor resection is associated with prolonged survival. The standard treatment uses conventional neuronavigation systems to increase extent of tumor resection. However, the quality of this form of neuronavigation decreases throughout surgery because of "brain shift". This is caused by edema, loss of cerebrospinal fluid and tumor resection. A new form of neuronavigation uses intraoperative MRI to compensate for brain shift, and to check for the presence of residual tumor that can be removed.

This study aims to compare the extent of glioblastoma resection between the standard treatment and intraoperative MRI.

ELIGIBILITY:
Inclusion Criteria:

* supratentorial brain tumor, on contrast enhanced dMRI suspected to be GBM
* indication for gross total resection (GTR) of the tumor
* age ≥18 years
* WHO Performance Scale ≤ 2
* ASA class ≤ 3
* adequate knowledge of the Dutch or French language
* informed consent

Exclusion Criteria:

* recurrent brain tumor
* multiple brain tumor localizations
* earlier skull radiotherapy
* earlier chemotherapy for GBM
* Chronic Kidney Disease or other renal function disorder
* known MR-contrast allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-02; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Difference in Residual tumor volume | <72h after surgery

SECONDARY OUTCOMES:
Complications, Clinical Performance, and Quality of Life | 3 months after surgery
Survival | 2 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Henk van Santbrink, MD, PhD, Principal Investigator — Maastricht University Medical Center; Didier Martin, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Liege; Koo van Overbeeke, MD, PhD, Study Chair — Maastricht University Medical Center
Locations (2):
- Centre Hospitalier Universitaire de Liege, Liège, Belgium
- Maastricht University Medical Center, Maastricht, Netherlands